CLINICAL TRIAL: NCT00584181
Title: High Resolution Computed Tomographic Evaluation of Airway Distensibility in Lung Transplant Recipients: A Pilot Study
Brief Title: High-resolution Computed Tomography (HRCT) Evaluation of Airway Distensibility in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 07-247
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Unspecified Complication of Lung Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung transplant recipients: Lung transplant recpients enrolled as study subjects will undergo pulmonary function tests (spirometry and lung volume measurements) and initial HRCT of chest. These subjects will receive nebulized ipratropium followed by pulmonary function tests (spirometry and lung volume measurements) and repeat HRCT.

SUMMARY:
Lung and heart-lung recipients at the University of Texas Medical Branch who have participated in the "Assessment of Cough Reflex in Lung Transplant Recipients" study who meet the specific study inclusion/exclusion criteria will have one study visit where they will undergo lung volume measurements, followed by high resolution CT scan of the lungs within 2 hours. After the initial CT scan, patients will be given a standard dose of Atrovent, followed thirty minutes later by repeat lung volume measurements and CT scan.

DETAILED DESCRIPTION:
Chest CT imaging will be obtained in the radiology department at UTMB. After the initial screening visit, subjects will visit the pulmonary function laboratory where they will undergo spirometry and measurement of lung volumes by whole body plethysmography. Within two hours of pulmonary function testing, subjects will undergo an initial HRCT scan. After the initial HRCT, subjects will inhale a standard dose of ipratropium bromide (0.5 mg) using a hand held nebulizer. Thirty minutes after ipratropium bromide administration, spirometry will be measured followed by a second HRCT scan.

Spirometry measurements will be performed in triplicate with the subjects in a seated position using a portable Koko spirometer (PDS, Louisville, CO). After the spirometry measurements, lung volumes will be measured in a body plethysmograph (MedGraphics, St. Paul, MN) with the subjects in a seated position with a nose clip. Subjects will be instructed to pant against the closed shutter at a frequency of 1-3 Hz. Lung volume measurements will be obtained prior to inital chest CT. Subjects will undergo high resolution computed tomography (HRCT) scanning within 30 minutes of initial lung volume measurements.

After the initial HRCT of the chest, subjects will inhale a dose of nebulized ipratropium bromide (0.5 mg) by standard nebulizer after which spirometry and lung volume measurements will be repeated in the pulmonary function laboratory. Spirometry and lung volume measurements will be performed in the same manner. Lung volume measurements will be obtained to account for changes in lung volumes after bronchodilator administration. Changes in lung volumes will be used to account for any changes noted on HRCT scans.

HRCT scanning will begin 6 cm above the top of the dome of the diaphragm, at TLC and moved caudally. Images will be reconstructed with the use of a high-spatial frequency (resolution) algorithm that enhanced edge detection, at a window level of -450 Hounsfield units and a window width of 1,350 Hounsfield units. We will consider the airway diameters after maximum bronchodilation with ipratropium to be a function principally of the structural characteristics of airways. The TLC measurements after ipratropium will be the best reflection of intrinsic structure. CT airway measurement analysis will be performed by VIDA Diagnostics. We have entered into a collaboration with VIDA Diagnostics that will allow accurate and reliable CT airway measurements. Subject's CT images obtained at UTMB will be deidentified and electronically transmitted to a research collaborator at VIDA Diagnostics located in Coralville, IA. The CT images will have a code assigned, known only to the PI. Using a proprietary software platform, airway measurements will be performed and the data electronically transmitted to the PI at UTMB.

ELIGIBILITY:
Inclusion Criteria:

* lung transplant recipients >18 years of age
* at least 12 months or greater from time of transplantation

Exclusion Criteria:

* hemodynamic instability
* hypoxemia
* pneumonia
* moderate or large pleural effusion
* clinical evidence of acute rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who participated in the "Assessment of Cough Reflex in Lung Transplant Recipients" study who meet the specific inclusion/exclusion criteria for this study
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2018-01-07 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Spirometry changes | Two hours (before and after inhalation of ipratropium)
  Assessment of changes in spirometry following inhalation of nebulized ipratropium

SECONDARY OUTCOMES:
Lung volumes | Two hours (before and after inhalation of ipratropium)
  Assessment of changes in total lung capacity, functional reserve capacity and inspiratory capacity following inhalation of nebulized ipratropium

OTHER OUTCOMES:
Radiographic changes in airway caliber | Two hours (before and after inhalation of ipratropium)
  Assessment of changes in airway caliber as determined by high resolution chest CT images following inhalation of nebulized ipratropium

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Duarte, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States